CLINICAL TRIAL: NCT03519412
Title: Pembrolizumab in MMR-Proficient Metastatic Colorectal Cancer Pharmacologically Primed to Trigger Dynamic Hypermutation Status
Brief Title: Pembrolizumab in MMR-Proficient Metastatic Colorectal Cancer Pharmacologically Primed to Trigger Hypermutation Status
Acronym: ARETHUSA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IFOM ETS - The AIRC Institute of Molecular Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFOM-CPT002/2018/PO001; 2018-001441-14 (EudraCT Number)
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Neoplasms; Microsatellite Instability
Keywords: DNA Mismatch Repair; Pembrolizumab
MeSH Terms: conditions — Colorectal Neoplasms; Microsatellite Instability | interventions — Temozolomide; Neoadjuvant Therapy; pembrolizumab; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MMR-proficient (MMRp) (Experimental): MGMT-IHC-negative, MGMT promoter methylation-positive patient population is selected for treatment with temozolomide (induction) orally until disease progression or unacceptable toxicity whichever comes first, followed by pembrolizumab IV if Tumor Mutational Burden post Temozolomide is > 20 Muts/Mb
  Interventions: Drug: temozolomide (induction),; Biological: pembrolizumab (treatment)
- MMR-deficient (MMRd) (Other): Patients receive Pembrolizumab (treatment) IV until disease progression or unacceptable toxicity or 35 cycles, whichever comes first
  Interventions: Biological: pembrolizumab (treatment)

INTERVENTIONS:
Drug: temozolomide (induction), — temozolomide is administered to MGMT promoter methylation-positive MMRp patients orally, once daily, at the dose of 150-200 mg/m2/day for 5 consecutive days of each treatment cycle A treatment cycle will comprise 5 days of temozolomide administration (Day 1 to 5) followed by 23 days of rest for a total of 28 days (4 weeks) period (dose-schedule: 150 mg/m2 day 1-5 q28),until disease progression or unacceptable toxicity whichever comes first.
  Other Names: methazolastone; Temodal; Temodar
  Arms: MMR-proficient (MMRp)
Biological: pembrolizumab (treatment) — pembrolizumab is administered to MGMT-IHC-negative, MGMT promoter methylation-positive MMRp patients with TMB>20 Mut/Mb after Temozolomide treatment, and to MMRd. Patients receive pembrolizumab IV , 200 mg Q3W, Day 1 of each 3 week cycle for maximum 35 cycles, until disease progression or unacceptable toxicity whichever comes first.
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
In this study, MMRd metastatic colorectal cancer (mCRC) patients who failed standard therapies will undergo treatment with pembrolizumab, while RAS-extended mutated MMR-proficient mCRC patients will be tested for o6-methylguanine-DNA-methyltransferase (MGMT) expression (IHC) and then for MGMT promoter methylation. MGMT IHC-negative, promoter methylation positive patients will be treated with temozolomide (TMZ). Patients progressing under temozolomide will be tested for tumor mutational burden (TMB) and proceed to pembrolizumab if TMB is > 20 mutations/Mb. The primary study hypothesis is that tumors with acquired resistance to temozolomide become hypermutated and are sensitive to pembrolizumab.

DETAILED DESCRIPTION:
Arethusa consists of three different phases - SCREENING Phase, PRIMING phase, and TRIAL Phase.

* SCREENING PHASE: MMR-Deficient (MMR-D) patients will proceed directly to TRIAL Phase (cohort D) to be treated with pembrolizumab. RAS mutant MMR-Proficient (MMR-P) patients, instead, are further tested for O6-methylguanine-DNA methyltransferase gene expression (MGMT) status in tissue (MGMT protein IHC and MGMT promoter methylation). MGMT IHC negative and promoter methylated patients will proceed to PRIMING phase.
* PRIMING PHASE: MMR-P patients showing negative MGMT protein and high levels of MGMT promoter methylation in tissues will receive TMZ therapy until progression. Two tumor biopsies will be taken prior to starting therapy and at progression to determine the mutational load. Patients with a mutational load < 20 mutations/megabase will go off-study. Patients with a mutational load >20 mutations/megabase, will proceed to trial phase no longer than week 5 post TMZ-ML.
* TRIAL PHASE: Eligible patients, i.e. MMRD patients (cohort D) and patients with a TMZ-ML > 20 mutations per megabase at TMZ-ML (cohort P), will be treated with pembrolizumab 200 mg administered as an intravenous infusion over 30 minutes every 3 weeks until disease progression, unacceptable toxicity, or up to 24 months in patients without disease progression.

ELIGIBILITY:
Inclusion Criteria:

Entry criteria for SCREENING Phase

1. Histologically confirmed diagnosis of metastatic colorectal cancer.
2. Documented RAS extended mutations in the archival sample (cohort P only).
3. ECOG performance status 0-1.
4. SCREENING phase informed consent signed.
5. Understanding and accepting the need for undergoing two tumor biopsies if eligible for PRIMING Phase.
6. Age ≥ 18 years.
7. Availability of all diagnostic FFPE blocks (primary tumor and or metastases), or at least 20 slides (primary tumor and/or metastases). Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
8. Normal organ functions.

Entry Criteria for PRIMING Phase

1. Fulfilment of all the SCREENING inclusion criteria;
2. PRIMING informed consent signed;
3. Confirming the willingness to undergo two tumor biopsies,
4. Acceptance that, if the mutational load determination is unfeasible for technical reasons (not enough tissue, substandard test performance, etc.), access to TRIAL phase will not be possible.
5. Imaging documented failure of previous standard CRC therapies including fluoropyrimidine, oxaliplatin, irinotecan plus or minus antiangiogenics agents (Bevacizumab, Aflibercept, Regorafenib, others).
6. At least one measurable tumor lesion as per RECIST v1.1. Lesions in previously irradiated areas or those that have received other loco-regional therapies (i.e.

   percutaneous ablation) should not be considered measurable unless there is clear documented evidence of progression of the lesion since therapy. Imaging must be performed maximum within 28 days prior to enrolment.
7. ECOG performance status 0 or 1;
8. Following results in the SCREENING Phase tests:

   * Proficient MMR status assessed by IHC or MSI-Low status defined by PCR (Bethesda panel);
   * Negative score for the MGMT protein expression IHC test;
   * Positive score for the MGMT promoter methylation performed on Tissue.
9. Women with childbearing potential should complete a pregnancy test and be willing to use highly effective contraceptive methods.
10. Normal organ functions.

Entry Criteria for TRIAL Phase

1. 1. Fulfilment of all the SCREENING inclusion criteria and Deficient MMR status (IHC) or MSI-High status (PCR) (cohort D only).
2. Fulfilment of all the SCREENING and PRIMING inclusion criteria (cohort P only).
3. TRIAL Phase informed consent signed (both cohorts).
4. Imaging documented PD to TMZ (cohort P only).
5. A mutational load value > 20 mutations/MB at TMZ-ML assay (cohort P only).
6. Imaging documented failure of previous standard CRC therapies including fluoropyrimidine, oxaliplatin, irinotecan plus or minus targeted agents (Bevacizumab, Aflibercept, Regorafenib, Cetuximab, Panitumumab, others) (cohort D only).
7. At least one measurable tumor lesion as per RECIST v1.1. Lesions in previously irradiated areas or those that have received other loco-regional therapies (i.e. percutaneous ablation) should not be considered measurable unless there is clear documented evidence of progression of the lesion since therapy. Imaging must be performed maximum within 28 days prior to enrolment (both cohorts).
8. Woman with childbearing potential should complete a pregnancy test and be willing to use highly effective contraceptive methods (both cohorts).
9. Normal organ functions. Blood specimens must be collected within 10 days prior to the start of study treatment (both cohorts).

Exclusion Criteria:

1. A woman of child bearing potential who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to allocation.

   1. Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.
   2. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Has received prior radiotherapy within 2 weeks of start of study treatment (with pembrolizumab). Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   a. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiological stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has severe hypersensitivity (≥Grade 3) to temozolomide and/or any of its excipients.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
13. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
14. Has an active infection requiring systemic therapy.
15. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required.
16. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
17. Has a known history of active TB (Bacillus Tuberculosis).
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
20. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Tumor assessments every 8-9 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Overall response rate (ORR) to pembrolizumab according to RECIST v1.1 and iRECIST

SECONDARY OUTCOMES:
Progression Free Survival | assessments every 8-9 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Progression Free Survival in MMRp pembrolizumab treated patients
Overall Survival | assessments every 8-9 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Overall Survival in MMRp pembrolizumab treated patients
Safety and Tolerability | assessments every 3 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Safety and Tolerability according to CTCAE version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Siena, MD, Study Chair — Grande ospedale metropolitano Niguarda; Silvia Marsoni, MD, Study Director — IFOM (Istituto FIRC di Oncologia Molecolare); Andrea Sartore bianchi, MD, Principal Investigator — Grande ospedale metropolitano Niguarda
Locations (4):
- Italy (4):
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori di Milano, Milan
  - Istituto Clinico Humanitas, Rozzano

REFERENCES:
- [Background] Amatu A, Sartore-Bianchi A, Moutinho C, Belotti A, Bencardino K, Chirico G, Cassingena A, Rusconi F, Esposito A, Nichelatti M, Esteller M, Siena S. Promoter CpG island hypermethylation of the DNA repair enzyme MGMT predicts clinical response to dacarbazine in a phase II study for metastatic colorectal cancer. Clin Cancer Res. 2013 Apr 15;19(8):2265-72. doi: 10.1158/1078-0432.CCR-12-3518. Epub 2013 Feb 19. PMID 23422094
- [Background] Amatu A, Barault L, Moutinho C, Cassingena A, Bencardino K, Ghezzi S, Palmeri L, Bonazzina E, Tosi F, Ricotta R, Cipani T, Crivori P, Gatto R, Chirico G, Marrapese G, Truini M, Bardelli A, Esteller M, Di Nicolantonio F, Sartore-Bianchi A, Siena S. Tumor MGMT promoter hypermethylation changes over time limit temozolomide efficacy in a phase II trial for metastatic colorectal cancer. Ann Oncol. 2016 Jun;27(6):1062-1067. doi: 10.1093/annonc/mdw071. Epub 2016 Feb 24. PMID 26916096
- [Background] Barault L, Amatu A, Bleeker FE, Moutinho C, Falcomata C, Fiano V, Cassingena A, Siravegna G, Milione M, Cassoni P, De Braud F, Ruda R, Soffietti R, Venesio T, Bardelli A, Wesseling P, de Witt Hamer P, Pietrantonio F, Siena S, Esteller M, Sartore-Bianchi A, Di Nicolantonio F. Digital PCR quantification of MGMT methylation refines prediction of clinical benefit from alkylating agents in glioblastoma and metastatic colorectal cancer. Ann Oncol. 2015 Sep;26(9):1994-1999. doi: 10.1093/annonc/mdv272. Epub 2015 Jun 25. PMID 26113646
- [Background] Bardelli A, Cahill DP, Lederer G, Speicher MR, Kinzler KW, Vogelstein B, Lengauer C. Carcinogen-specific induction of genetic instability. Proc Natl Acad Sci U S A. 2001 May 8;98(10):5770-5. doi: 10.1073/pnas.081082898. Epub 2001 Apr 10. PMID 11296254
- [Background] Germano G, Lamba S, Rospo G, Barault L, Magri A, Maione F, Russo M, Crisafulli G, Bartolini A, Lerda G, Siravegna G, Mussolin B, Frapolli R, Montone M, Morano F, de Braud F, Amirouchene-Angelozzi N, Marsoni S, D'Incalci M, Orlandi A, Giraudo E, Sartore-Bianchi A, Siena S, Pietrantonio F, Di Nicolantonio F, Bardelli A. Inactivation of DNA repair triggers neoantigen generation and impairs tumour growth. Nature. 2017 Dec 7;552(7683):116-120. doi: 10.1038/nature24673. Epub 2017 Nov 29. PMID 29186113
- [Derived] Willis JA, Overman MJ. Inducing Hypermutability to Promote Anti-PD-1 Therapy Response. Cancer Discov. 2022 Jul 6;12(7):1612-1614. doi: 10.1158/2159-8290.CD-22-0492. PMID 35791694